CLINICAL TRIAL: NCT04206670
Title: Developing and Evaluating In-Home Supportive Technology for Caregivers of People With Dementia and Mild Cognitive Impairment
Brief Title: In-Home Technology for Caregivers of People With Dementia and Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: People Power Company (Industry); National Institute on Aging (NIA) (NIH); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Robert Levenson, Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R44AG059458-03 (NIH); R44AG059458 (NIH)
Record Dates: First submitted 2019-12-10; First posted 2019-12-20 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Dementia; Mild Cognitive Impairment; Alzheimer Disease
Keywords: Caregivers; Dementia; Mild Cognitive Impairment; In-Home Technology; Alzheimer Disease
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Alzheimer Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Participants are randomly assigned to treatment arms by People Power. All participants complete the same questionnaires at the same intervals. University of California, Berkeley investigators are blind as to participants' treatment arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Home Technology System (Experimental): Participants will receive and install the full system (sensors for entry, activity, temperature, water leak; voice control; digital display; local router) in their homes. Remote assistance will be provided to help with the installation. Sensors, warnings, messaging, and social networking features will be activated remotely. Participation will extend over a six month period with questionnaires (e.g., health and well-being) administered 3 times (at the time of installation and every 3 months thereafter).
  Interventions: Device: In-Home Technology System and Questionnaires
- Waiting Control (Other): Participants will be assigned a date for receiving and installing the full system (sensors for entry, activity, temperature, water leak; voice control; digital display; local router) six months after they enter the study. During that six-month period, questionnaires (e.g., health and well-being) will be administered 3 times (at the start of the study and every 3 months thereafter). At the end of the six-month period, participants will receive and install the full system (sensors for entry, activity, temperature, water leak; voice control; digital display; local router) in their homes. Remote assistance will be provided to help with the installation. Sensors, warnings, messaging, and social networking features will be activated remotely. Participation will extend over an additional six-month period with questionnaires (e.g., health and well-being) administered 2 times (every 3 months following installation).
  Interventions: Device: Waiting Control In-Home Technology System and Questionnaires

INTERVENTIONS:
Device: In-Home Technology System and Questionnaires — Participants self-install the in-home technology system in their homes after enrollment in the study (i.e., consent procedures and initial questionnaire). Intelligent bots monitor the in-home sensors, learn typical patterns, and provide caregivers with text messages via cell phone and alerts via the tablet when worrisome behaviors occur. Social contact is encouraged using caregiver resources and a trusted circle of friends and family who are encouraged to stay in contact with the caregiver and person with dementia or mild cognitive impairment.
  Arms: In-Home Technology System
Device: Waiting Control In-Home Technology System and Questionnaires — Participants self-install the in-home technology system in their homes six months after their enrollment in the study (i.e., consent procedures and initial questionnaire). Intelligent bots monitor the in-home sensors, learn typical patterns, and provide caregivers with text messages via cell phone and alerts via the tablet when worrisome behaviors occur. Social contact is encouraged using caregiver resources and a trusted circle of friends and family who are encouraged to stay in contact with the caregiver and person with dementia or mild cognitive impairment.
  Arms: Waiting Control

SUMMARY:
This study aims to develop and evaluate new in-home supportive technology that is designed to alleviate anxiety, burden, and loneliness in spousal and familial caregivers of individuals with Alzheimer's disease, other dementias, or mild cognitive impairment.

DETAILED DESCRIPTION:
This study aims to develop, refine, and evaluate a new hardware/software system designed to integrate in-home sensors and devices, Internet-of-Things technologies (i.e., devices that can be controlled and communicated with via the internet), and social networking to create a more safe and supportive home environment for caregivers and people who have Alzheimer's disease, other dementias, or mild cognitive impairment. The system monitors troublesome behaviors in people with dementia or mild cognitive impairment (e.g., wandering), and targets mechanisms (e.g., worry, social isolation) thought to link behavioral symptoms in people with dementia or mild cognitive impairment with adverse caregiver outcomes (declines in health and well-being). The system is designed to minimize demands on caregivers' limited time and energy and to provide a platform for data collection that can be used by researchers and care professionals.

Hypotheses:

1. Caregivers in the full operation condition will have fewer negative effects of caregiving (lower burden, better mental and physical health, higher well-being) than those in the control condition.
2. Greater use of the social networking features of the system will be associated with fewer caregiver depressive symptoms.
3. Greater utilization of the home safety features of the system will be associated with fewer caregiver anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers are fluent/literate in English
* Caregivers currently reside with spouse/family member who has received a diagnosis of Alzheimer's disease, other dementias, or mild cognitive impairment
* Caregivers primarily use a smartphone (e.g., iPhone, Android)
* Caregiver has wireless internet in home

Exclusion Criteria:

* Caregivers providing care for individuals with known non-neurodegenerative conditions affecting behavior and cognition
* Caregivers providing care for individuals with longstanding Axis I psychiatric disorder
* Caregivers providing care for individuals with metabolic disorder or major organ dysfunction
* Caregivers providing care for individuals with alcohol abuse or dependence (within 5 years of dementia onset)
* Caregivers providing care for individuals with head trauma with loss of consciousness greater than 30 minutes
* Caregivers providing care for individuals with contraindications to MRI imaging
* Caregivers providing care for individuals with large confluent white matter lesions
* Caregivers providing care for individuals with significant systemic medical illness
* Caregivers providing care for individuals who use a medication likely to affect central nervous system functions adversely

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Levenson, Ph.D., Study Director — University of California, Berkeley
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Because health and other protected data are involved, we need to consult with our institutional review board and other collaborators concerning which data can be shared.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Chen KH, Wells JL, Otero MC, Lwi SJ, Haase CM, Levenson RW. Greater Experience of Negative Non-Target Emotions by Patients with Neurodegenerative Diseases Is Related to Lower Emotional Well-Being in Caregivers. Dement Geriatr Cogn Disord. 2017;44(5-6):245-255. doi: 10.1159/000481132. Epub 2017 Dec 8. PMID 29216633
- [Background] Lwi SJ, Ford BQ, Casey JJ, Miller BL, Levenson RW. Poor caregiver mental health predicts mortality of patients with neurodegenerative disease. Proc Natl Acad Sci U S A. 2017 Jul 11;114(28):7319-7324. doi: 10.1073/pnas.1701597114. Epub 2017 Jun 27. PMID 28655841
- [Background] Otero MC, Levenson RW. Lower Visual Avoidance in Dementia Patients Is Associated with Greater Psychological Distress in Caregivers. Dement Geriatr Cogn Disord. 2017;43(5-6):247-258. doi: 10.1159/000468146. Epub 2017 Apr 11. PMID 28395276
- [Background] Brown CL, Lwi SJ, Goodkind MS, Rankin KP, Merrilees J, Miller BL, Levenson RW. Empathic Accuracy Deficits in Patients with Neurodegenerative Disease: Association with Caregiver Depression. Am J Geriatr Psychiatry. 2018 Apr;26(4):484-493. doi: 10.1016/j.jagp.2017.10.012. Epub 2017 Dec 27. PMID 29289452
- [Derived] Bullard BM, Brown CL, Scheffer JA, Toledo AB, Levenson RW. Emotion Regulation Strategies and Mental Health in Dementia Caregivers: The Moderating Role of Gender. Dement Geriatr Cogn Disord. 2024;53(3):128-134. doi: 10.1159/000538398. Epub 2024 Apr 22. PMID 38537622
- See also: Presence Caregiver Research Website — https://research.presencefamily.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note that outcomes are only assessed regarding caregiver health and well-being. Patients did not provide any information; therefore, all information reported for demographics and measures is only regarding caregivers.
Groups:
- Waiting Control: Participants will be assigned to receive and install the full system (sensors for entry, activity, temperature, water leak; voice control; digital display; local router) after they enter the study. During a 6-month period, questionnaires (e.g., health and well-being) will be administered 3 times (at the start of the study and every 3 months thereafter). Remote assistance will be provided to help with the installation. Sensors, warnings, messaging, and social networking features will be activated remotely. Participation will extend over an additional 6-month period with questionnaires (e.g., health and well-being) administered 2 times (every 3 months following installation).
  Waiting Control In-Home Technology System and Questionnaires: Participants self-install the in-home technology system in their homes six months after their enrollment in the study (i.e., consent procedures and initial questionnaire). Intelligent bots monitor the in-home sensors, learn typical patterns, and provide caregivers with text messages via cell phone and alerts via the tablet when worrisome behaviors occur. Social contact is encouraged using caregiver resources and a trusted circle of friends and family who are encouraged to stay in contact with the caregiver and person with dementia or mild cognitive impairment.
Period: Overall Study
Arm/Group | In-Home Technology System | Waiting Control
Started | 148 | 68
Completed | 124 | 65
Not Completed | 24 | 3

BASELINE CHARACTERISTICS:
Groups:
- In-Home Technology System; Waiting Control: Participants (N=300) will receive and install the full system (sensors for entry, activity, temperature, water leak; voice control; digital display; local router) in their homes. Remote assistance will be provided to help with the installation. Sensors, warnings, messaging, and social networking features will be activated remotely. Participation will extend over a six month period with questionnaires (e.g., health and well-being) administered 3 times (at the time of installation and every 3 months thereafter).
  In-Home Technology System and Questionnaires: Participants self-install the in-home technology system in their homes after enrollment in the study (i.e., consent procedures and initial questionnaire). Intelligent bots monitor the in-home sensors, learn typical patterns, and provide caregivers with text messages via cell phone and alerts via the tablet when worrisome behaviors occur. Social contact is encouraged using caregiver resources and a trusted circle of friends and family who are encouraged to stay in contact with the caregiver and person with dementia or mild cognitive impairment.
- Total: Total of all reporting groups
Arm/Group | In-Home Technology System | Waiting Control | Total
Number analyzed (Participants) | 148 | 68 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (11.8) | 64.6 (9.8) | 63.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 51 | 141
  Male | 58 | 17 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 8 | 3 | 11
  East Asian, South Asian, Southeast Asian, or Indian American | 9 | 4 | 13
  Latino or Hispanic American | 8 | 4 | 12
  Native Hawaiian or Pacific Islander | 1 | 1 | 2
  Non-Hispanic White or European American | 108 | 51 | 159
  Other | 14 | 5 | 19
Beck Anxiety Inventory [Mean (Standard Deviation); unit: units on a scale] | 7.36 (8.23) | 9.46 (7.12) | 8.02 (7.94)
Zarit Burden Inventory [Mean (Standard Deviation); unit: units on a scale] | 20.04 (8.71) | 21.35 (8.13) | 20.45 (8.53)
Satisfaction with Life [Mean (Standard Deviation); unit: units on a scale] | 20.99 (7.24) | 18.81 (6.85) | 20.30 (7.18)
Center for Epidemiologic Studies Depression Scale [Mean (Standard Deviation); unit: units on a scale] | 15.14 (10.04) | 17.90 (10.44) | 16.01 (10.22)

OUTCOME MEASURES:

1. Primary Outcome: 3 Months Assessment for Center for Epidemiological Studies Depression Scale (CES-D)
Description: Questionnaire to measure depression (Radloff, 1977). 20 items are rated on a 0-3 scale and summed (range = 0-60). There are no subscales. Higher scores represent worse outcomes. The clinical cut-off is usually set at a score of 16.
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Waiting Control
Number analyzed (Participants) | 125 | 61
units on a scale | 16.05 (10.30) | 18.39 (10.27)

2. Primary Outcome: 6 Months Assessment for Center for Epidemiological Studies Depression Scale (CES-D)
Description: as for outcome 1
Time Frame: 6 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Waiting Control: Participants (N=100) will be assigned to receive and install the full system (sensors for entry, activity, temperature, water leak; voice control; digital display; local router) after they enter the study. During a 6-month period, questionnaires (e.g., health and well-being) will be administered 3 times (at the start of the study and every 3 months thereafter). Remote assistance will be provided to help with the installation. Sensors, warnings, messaging, and social networking features will be activated remotely. Participation will extend over an additional 6-month period with questionnaires (e.g., health and well-being) administered 2 times (every 3 months following installation).
  Waiting Control In-Home Technology System and Questionnaires: Participants self-install the in-home technology system in their homes six months after their enrollment in the study (i.e., consent procedures and initial questionnaire). Intelligent bots monitor the in-home sensors, learn typical patterns, and provide caregivers with text messages via cell phone and alerts via the tablet when worrisome behaviors occur. Social contact is encouraged using caregiver resources and a trusted circle of friends and family who are encouraged to stay in contact with the caregiver and person with dementia or mild cognitive impairment.
Arm/Group | In-Home Technology System | Waiting Control
Number analyzed (Participants) | 122 | 64
units on a scale | 15.98 (11.61) | 17.17 (9.55)

3. Primary Outcome: 3 Months Assessment for Zarit Burden Interview-Short Form
Description: Questionnaire to measure caregiver burden (Zarit, Reever, & Bach-Peterson, 1980). 12 items are rated on 0-4 scale. Range: 0-48. No subscales. Higher scores represent worse outcomes.
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Waiting Control
Number analyzed (Participants) | 121 | 61
units on a scale | 20.40 (9.19) | 21.31 (8.63)

4. Primary Outcome: 6 Months Assessment for Zarit Burden Interview-Short Form
Description: as for outcome 3
Time Frame: 6 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Waiting Control
Number analyzed (Participants) | 116 | 61
units on a scale | 20.93 (9.17) | 21.87 (8.86)

5. Primary Outcome: 3 Months Assessment for Beck Anxiety Inventory (BAI)
Description: Questionnaire to measure anxiety (Beck, Epstein, Brown, & Steer, 1988). 20 items are rated on a 0-3 scale and summed (range= 0-60). Higher scores indicate worse outcomes. There are no subscales. A score greater than 36 is considered to be clinically significant.
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Waiting Control
Number analyzed (Participants) | 125 | 63
units on a scale | 8.06 (7.71) | 9.29 (7.55)

6. Primary Outcome: 6 Months Assessment for Beck Anxiety Inventory (BAI)
Description: as for outcome 5
Time Frame: 6 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Waiting Control
Number analyzed (Participants) | 122 | 65
units on a scale | 7.81 (8.44) | 8.71 (6.53)

7. Primary Outcome: 3 Months Assessment for Satisfaction With Life Scale
Description: Questionnaire measuring overall life satisfaction and well-being (Diener, Emmons, Larsen, & Griffin, 1985). 5 items scored on a 1-7 scale and summed (Range = 5-35). Lower scores indicate worse outcomes. A score of 20 is considered neutral with higher scores considered increasingly more satisfied and lower scores considered increasingly more dissatisfied.
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Waiting Control
Number analyzed (Participants) | 125 | 63
units on a scale | 21.26 (6.96) | 18.68 (7.11)

8. Primary Outcome: 6 Months Assessment for Satisfaction With Life Scale
Description: as for outcome 7
Time Frame: 6 months after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | In-Home Technology System | Waiting Control
Number analyzed (Participants) | 121 | 65
units on a scale | 21.28 (7.51) | 18.66 (7.06)

ADVERSE EVENTS:
Time Frame: Baseline to 6 months
Arm/Group | In-Home Technology System | Waiting Control
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/68
Other Adverse Events (participants affected / at risk) | 0/148 | 0/68

LIMITATIONS AND CAVEATS:
The study intended to recruit 400 participants, however at the start of enrollment, COVID-19 shutdowns occurred and caregivers were less likely to enroll in the study because they were at home (i.e., not out in public) more often, thus not needing to remotely monitor the individuals that they were providing care for. Thus the final number of installations was 216. Due to selective attrition the final active control ratio was approximately 2:1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT04206670/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT04206670/SAP_001.pdf